CLINICAL TRIAL: NCT07158801
Title: A Web-based Single Session Intervention to Reduce Caregiver Distress and Accommodation in Socioeconomically Diverse Caregivers of OCD Patients
Brief Title: Project EMPOWER-OCD
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Jenna Sung, PhD, Assistant Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 8178E
Record Dates: First submitted 2025-09-03; First posted 2025-09-08 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Parental Accommodation; Obsessive-Compulsive Disorder; Caregiving; Single Session Interventions
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Project EMPOWER-OCD (Experimental): Project EMPOWER-OCD is a web-based intervention for caregivers that takes about 20-25 minutes to complete that reduces accommodation.
  Interventions: Behavioral: Project EMPOWER-OCD
- Project CARE (Active Comparator): This active psychoeducation-based SSI will provide general information on caregiving and caregiver mental health.
  Interventions: Behavioral: Project CARE

INTERVENTIONS:
Behavioral: Project EMPOWER-OCD — Project EMPOWER-OCD is a web-based intervention for caregivers that takes about 20-25 minutes to complete that reduces accommodation. The program is drawing from an empirically supported intervention, Project EMPOWER, and will be adapted for the OCD population pending stakeholder input during phase 1 and include 5 elements: (1) an introduction to the program's rationale; (2) psychoeducation around OCD-driven avoidance, along with how caregiver accommodation can inadvertently maintain these avoidance patterns; (3) information on how caregivers can better identify patterns of avoidance, validate, and encourage approach behaviors instead; (4) creation of an "action plan" to promote approach behavior and reducing avoidance; (5) a vignette exercise in which caregivers read about another case and provide possible solutions based on what they learned. Resources for finding mental health treatment for OCD are presented at the end.
  Arms: Project EMPOWER-OCD
Behavioral: Project CARE — To evaluate the effects of Project EMPOWER-OCD, we will compare it to an active psychoeducation-based SSI that provides general information on caregiving and caregiver mental health. The intervention includes 5 elements that mirror Project EMPOWER: (1) introduction to the rationale for the program; (2) introduce the concept of caregiving across relationships and situations; (3) present broad information on typical development processes; (4) helping caregivers identify their own role and reflect on how caregiving looks like in their life (5) vignette exercise where caregivers identify caregiving roles, prompting reflection on roles. This active comparator intentionally does not include any psychoeducational components explicitly designed to reduce accommodation of anxiety, OCD, and its related disorders.
  Arms: Project CARE

SUMMARY:
This research study aims to adapt and evaluate the acceptability and effectiveness of Project EMPOWER-OCD for socioeconomically diverse caregivers of patients with OCD. Designed to reduce obstacles (e.g. months long time commitment, high cost, transportation) to treatment that caregivers may be particularly prone to, project EMPOWER-OCD will provide targeted intervention of accommodation - a well-established, potentially modifiable risk factor for child anxiety, OCD, and its related disorders - in a single, self-guided session via an online format.

DETAILED DESCRIPTION:
The need for accessible, effective interventions for child OCD that meet the needs of financially insecure families can be addressed via mechanism-targeted single session interventions (SSIs). Unlike the dominant models of brick-and-mortar clinic based, multi-week psychotherapy, SSIs involve intentional, single visit or interaction with a clinic, provider, or self-guided program. To date, SSIs have prevented and reduced child psychopathology across numerous trials . Given that the modal number of therapy sessions completed across all care settings is one, SSIs leverage these one-time interactions to complement -rather than replace -the existing mental health care models to help address long-standing, multi-level barriers to care (e.g., lack of providers, long waitlists, and family's ability to attend multi-sessions).

In SSI development, it is critical to identify target mechanisms to optimize the likelihood of spurring clinical change in a short period of time. One way caregivers get further entangled in the webs of OCD is accommodation, which refers to changes in caregiving behaviors or routines that facilitate or maintain their child's avoidance or anxiety. Examples include modifying family routines (i.e. adjusting work schedules to ensure the child has enough time to complete rituals) or directly participating in a patient's avoidance strategies (i.e. repeatedly washing objects on behalf of a patient who has contamination fears). Accommodation reduces the patient's short-term distress but inadvertently maintains their long-term avoidance. High levels of family accommodation have consistently predicted the maintenance and severity of OCD problems. Moreover, as accommodation involves the act of doing more to alleviate the patient's distress in the short term, reducing this common caregiving behavior gives caregivers the permission to do less - not only removing a common maintenance factor of OCD, but also decreasing caregiver burden and stress, ultimately improving family well-being. Project EMPOWER is a self-administered SSI that has been evaluated in previous trials to successfully reduce accommodation in caregivers of anxious children.

This research study aims to adapt and evaluate the acceptability and effectiveness of Project EMPOWER-OCD for socioeconomically diverse caregivers of patients with OCD. Designed to reduce obstacles (e.g. months long time commitment, high cost, transportation) to treatment that caregivers may be particularly prone to, project EMPOWER-OCD will provide targeted intervention of accommodation - a well-established, potentially modifiable risk factor for child anxiety, OCD, and its related disorders - in a single, self-guided session via an online format. SSIs have been shown to produce benefits across a range of mental health conditions and access to the intervention may provide potential benefits to their emotional health and family functioning. There are no known risks to participate in this study

ELIGIBILITY:
Inclusion Criteria:

* be a caregiver for at least one individual with OCD, defined as living in the same household and providing daily care
* be 18 years old or older
* the individual they are caring for have clinically significant OCD symptoms, indicated by a score a 16 or above on the self-reported Children's Yale-Brown Obsessive Compulsive Scale - Parent Report (CY-BOCS-PR)
* speak, read, and write English
* not be in concurrent family-based CBT treatment for the patient's OCD.

Exclusion Criteria:

* does not speak English
* younger than 18 years old
* participation in concurrent family-based CBT treatment for the patient's OCD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Family Accommodation Scale | Change from baseline, 2-week follow-up, 4-week follow-up
  19-item measure designed to assess the child's OCD symptoms and the extent to which a caregiver accommodates a child's OCD symptoms. Only the part two of the measure will be used to get the report of family member's responses to OCD. Items are rated from 0 (never) to 4 (every day). Total sum score ranges from 0 to 76 with higher scores indicating more frequent parental accommodation.
Children's Yale-Brown Obsessive Compulsive Scale | Change from baseline, 2-week follow-up, 4-week follow-up
  A two-part measure with a checklist of common obsessions and compulsions as well as a 10-item part that asks participants to report on the severity of their child's OCD rated on a 0 (none) to 4 (extreme) scale. Total sum score ranges from 0 to 40 with higher scores indicating higher symptom severity.

SECONDARY OUTCOMES:
Parental Stress Scale | Change from baseline, 2-week follow-up, 4-week follow-up
  An 18-item measure of caregiving stress levels, rated on a scale of 1 (strongly disagree) to a 5 (strongly agree) scale on their perceived positive and negative experience of being a caregiver
Program Feedback Scale | Immediately after the SSI
  The program feedback scale asks participants to rate 7 statements regarding acceptability and feasibility; note whether they would recommend this activity to others; and share what they liked and would change about the SSI. The 7 statements are rated from 0 (Really Disagree) to 5 (Really Agree). Total score ranges from 0 to 35, with higher scores indicating a more positive program evaluation.
Perceived pre-to-post SSI change | Immediately after the SSI
  a 2-item measure assesses participants' perceived change in their ability to help their children manage distressing situations from pre- to post-SSI: "compared to before you completed this program, how prepared do you feel to help your child manage distressing situations?" Participants in both groups will rate this question on a 5- point scale of 1 (much less able to help) to 5 (much more able to help).

OTHER OUTCOMES:
Consumer Financial Protection Bureau Financial Well-Being Scale | Baseline
  The CFPB Financial Well-Being Scale measures financial well-being as it relates to control over finances, capacity to absorb financial shock, and having the financial freedom to enjoy life. Parents are asked to answer 10 questions on a 0 to 4 Likert scale to generate a sum score, which is converted into a standardized score. Scores range from 14 to 95 with higher scores indicating a higher level of measure financial well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Access Criteria: Please contact the study PI for access